CLINICAL TRIAL: NCT06236685
Title: Optimizing the Assessment of Mechanical Ventilation by Integrating Advanced Monitoring Techniques
Brief Title: Optimizing the Assessment of Mechanical Ventilation by Integrating Advanced Monitoring Techniques [AVIM]
Acronym: AVIM
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Czech Technical University in Prague (Other)
Collaborators: Military University Hospital, Prague (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: AVIM
Record Dates: First submitted 2024-01-24; First posted 2024-02-01 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Mechanical Ventilation Complication; Ventilator-Induced Lung Injury
Keywords: electrical impedance tomography; expiratory time constant; mechanical energy; lung protective ventilation; ventilator-induced lung injury; expiratory flow; inspiratory hold maneuver
MeSH Terms: conditions — Ventilator-Induced Lung Injury

STUDY DESIGN:
Intervention Model Description: The study will be conducted on patients provided with mechanical ventilation either on intensive care units or during anesthesia. Extended monitoring of ventilation, including electric impedance tomography and esophageal pressure readings will be applied.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- General anesthesia (Experimental): Patients undergoing general anesthesia with mechanical ventilation will be monitored by electrical impedance tomography in addition to standard monitoring. Moreover, esophageal pressure catheter will be used in cases where indicated by clinician or in case of an indication of nasogastric tube, as esophageal pressure can be measured by a combined catheter.
  Interventions: Device: Electric impedance tomography
- Intensive Care Unit (Experimental): Patients ventilated in the ICU for various reasons will receive standard care, including advanced monitoring of mechanical ventilation.
  Interventions: Device: Electric impedance tomography

INTERVENTIONS:
Device: Electric impedance tomography — EIT is rarely used during general anesthesia for standard procedures. In the anesthesia arm, all patients will be monitored by EIT.
  Other Names: EIT

SUMMARY:
The aim of this study is to collect synchronized data from multiple monitoring techniques of mechanical ventilation (pressure/flow waves from the ventilator, electrical impedance tomography - EIT, esophageal pressure, capnography) in patients ventilated either on intensive care units or during anesthesia and evaluate the data by detailed mathematical analysis, to test three hypotheses:

1. Various published methods of calculation of the expiratory time constant provide different results in most cases.
2. Inhomogeneous ventilation (as described by EIT) affects the form of the expiratory flow curve and thus the calculated expiratory time constants.
3. The calculation of mechanical energy transferred to the lungs is affected by the chosen technique and length of the inspiratory pause maneuver.

This study does not test any new or non-standard methods and does not in any way interfere with the course of treatment indicated by the clinician, apart from extending the monitoring techniques.

DETAILED DESCRIPTION:
Mechanical ventilation is known to cause various complications, generally known as ventilator induced lung injury. Thus, detailed monitoring is essential. However, data interpretation is complicated in clinical practice. The investigators aim to collect synchronized data from multiple monitoring techniques of mechanical ventilation (pressure/flow waves from the ventilator, electrical impedance tomography - EIT, esophageal pressure, capnography) in patients ventilated either on intensive care units or during anesthesia and evaluate the data by detailed mathematical analysis. The results will be used to explore the complexity of seemingly simple and often used calculations describing the course of mechanical ventilation - mostly the expiratory time constant and amount of mechanical energy transferred to the lungs. The investigators primarily aim to test three hypotheses:

1. Various published methods of calculation of the expiratory time constant provide different results in most cases.
2. Inhomogeneous ventilation (as described by EIT) affects the form of the expiratory flow curve and thus the calculated expiratory time constants.
3. The calculation of mechanical energy transferred to the lungs is affected by the chosen technique and length of the inspiratory pause maneuver.

For this, the investigators plan to recruit 50 patients undergoing general anesthesia with controlled mechanical ventilation and 50 patients hospitalized on intensive care units. Monitoring of those patients will be protocolized and will in all cases include pressure/flow monitoring of the mechanical ventilator, capnography, and electrical impedance tomography. Esophageal pressure monitoring will be introduced where indicated by the clinician or where nasogastric tube insertion will be indicated (as the pressure can be measured by a combined catheter).

This study thus does not test any new or non-standard methods and does not in any way interfere with the course of treatment indicated by the clinician, apart from extending the monitoring techniques. Patient data will be anonymized and all the enrolled patients or their families will sign an informed consent as agreed by the ethical committee of our hospital.

ELIGIBILITY:
Inclusion Criteria:

* mechanical ventilation for anesthesia or in intensive care unit

Exclusion Criteria:

* disagreement with enrollment or incapacity to understand the patient information leaflet
* contraindications to electric impedance tomography (skin lesions in the place of electrode placement etc.)
* necessity to use a defined ventilator setting outside the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-04-22 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Expiratory time constant | 2 minutes after an intervention or a change in the ventilator settings
  Time [in seconds], in which the lungs exhale 63% of the total volume.
Mechanical energy transferred to the lungs | 2 minutes after an intervention or a change in the ventilator settings
  Mechanical energy (alternatively referred to as mechanical work) [in Joules] is the energy delivered to the respiratory system during a single inspiration cycle.

OTHER OUTCOMES:
Regional signals of electrical impedance tomography | 2 minutes after an intervention or a change in the ventilator settings
  Changes of regional signals of electrical impedance tomography throughout the respiratory cycle correspond to changes in lung aeration.

CONTACTS AND LOCATIONS:
Overall Officials: Karel Roubík, prof., Study Director — Czech Technical University
Locations (1):
- Military University Hospital, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No
If any particularly interesting cases arise, the investigators plan to share the individual monitoring data together with the study protocol as anonymized case studies, either published or upon request to other researchers.

REFERENCES:
- [Background] Karagiannidis C, Waldmann AD, Roka PL, Schreiber T, Strassmann S, Windisch W, Bohm SH. Regional expiratory time constants in severe respiratory failure estimated by electrical impedance tomography: a feasibility study. Crit Care. 2018 Sep 21;22(1):221. doi: 10.1186/s13054-018-2137-3. PMID 30236123
- [Background] Brunner JX, Laubscher TP, Banner MJ, Iotti G, Braschi A. Simple method to measure total expiratory time constant based on the passive expiratory flow-volume curve. Crit Care Med. 1995 Jun;23(6):1117-22. doi: 10.1097/00003246-199506000-00019. PMID 7774225
- [Background] Candik P, Rybar D, Depta F, Sabol F, Kolesar A, Galkova K, Torok P, Donicova V, Imrecze S, Nosal M, Donic V. Relationship between dynamic expiratory time constant tau(edyn) and parameters of breathing cycle in pressure support ventilation mode. Physiol Res. 2018 Dec 18;67(6):875-879. doi: 10.33549/physiolres.933750. Epub 2018 Sep 11. PMID 30204464
- [Background] Henderson WR, Molgat-Seon Y, Vos W, Lipson R, Ferreira F, Kirby M, Holsbeke CV, Dominelli PB, Griesdale DE, Sekhon M, Coxson HO, Mayo J, Sheel AW. Functional respiratory imaging, regional strain, and expiratory time constants at three levels of positive end expiratory pressure in an ex vivo pig model. Physiol Rep. 2016 Dec;4(23):e13059. doi: 10.14814/phy2.13059. PMID 27923979
- [Background] Vogt B, Pulletz S, Elke G, Zhao Z, Zabel P, Weiler N, Frerichs I. Spatial and temporal heterogeneity of regional lung ventilation determined by electrical impedance tomography during pulmonary function testing. J Appl Physiol (1985). 2012 Oct;113(7):1154-61. doi: 10.1152/japplphysiol.01630.2011. Epub 2012 Aug 16. PMID 22898553